CLINICAL TRIAL: NCT04050787
Title: Study on Laparoscopic No. 10 Lymph Node Dissection With Preservation of Spleen for Advanced Middle or Upper Third Gastric Cancer
Brief Title: Spleen-Preserving No. 10 Lymph Node Dissection in Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jian Suo (Other)
Responsible Party: Sponsor-Investigator, Jian Suo, professor, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No. 10 Lymph Node Dissection
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Overall Survival

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D2 Lymphadenectomy including No. 10 (Experimental): lymphadenectomy including spleen-preserving No. 10 lymph node dissection will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: D2 Lymphadenectomy including No. 10
- D2 lymphadenectomy excluding No. 10 (Active Comparator): Laparoscopic total gastrectomy with D2 lymphadenectomy but without No. 10 lymph node dissection will be performed for the treatment of patients assigned to this group
  Interventions: Procedure: D2 lymphadenectomy excluding No. 10

INTERVENTIONS:
Procedure: D2 Lymphadenectomy including No. 10 — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, Laparoscopic total gastrectomy with D2 lymphadenectomy including spleen-Preserving No. 10 Lymph Node Dissection will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy
  Arms: D2 Lymphadenectomy including No. 10
Procedure: D2 lymphadenectomy excluding No. 10 — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, Laparoscopic total gastrectomy with D2 lymphadenectomy excluding spleen-Preserving No. 10 Lymph Node Dissection will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience and anastomotic procedure is performed extracorporeally using a mini-laparotomy
  Arms: D2 lymphadenectomy excluding No. 10

SUMMARY:
This study is to conduct a randomized controlled trial of two kinds of radical gastrectomy for patients with proximal gastric cancer. One is laparoscopic D2 radical total gastrectomy combined with spleen-preserving No.10 lymph node dissection , another one is laparoscopic D2 radical total gastrectomy without clearing the No. 10 lymph nodes of the spleen. We explore the effect of the two procedures on the survival of patients, as well as the surgical complications associated with the two procedures, the number of lymph node dissection, the operation time and the amount of intraoperative blood loss. Furthermore, we also want to discuss the application value of laparoscopic lymph node dissection for spleen preservation in radical gastrectomy for proximal gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 80 years
2. Primary distal gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. cT2-4a, N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
4. No distant metastasis is observed. And the spleen, pancreas or other adjacent organs are not involved by the tumor.
5. Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
6. American Society of Anesthesiology score (ASA) class I, II, or III
7. Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
5. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
6. History of other malignant disease within past five years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within past six months
9. History of cerebrovascular accident within past six months
10. History of continuous systematic administration of corticosteroids within one month
11. Requirement of simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. FEV1<50% of predicted values

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-21 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | 36 months

SECONDARY OUTCOMES:
Morbidity | 30 days; 36 months
  The early postoperative complication are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
3-year overall survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
The number of lymph node dissection | 1 day
The number of positive lymph nodes | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jian Suo, Study Chair — Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No